# **Statistical Analysis Plan**

Clinical trial protocol title: Randomized, placebo-controlled trial of YF476, a gastrin receptor antagonist, in Barrett's esophagus HMR code: 10-505 T-016 Sponsor code: EudraCT no: 2014-002418-22 CRO details: Hammersmith Medicines Research Cumberland Avenue London NW10 7EW Sponsor details: Trio Medicines Ltd Hammersmith Medicines Research Cumberland Avenue London **NW10 7EW** Issued: 10 January 2019 Version: 1 Based on: Protocol version 24, 26 April 2018 Number of pages: 46 Prepared by: Stephen Sah

# **Table of contents**

| 1 | LIST | OF ABBREVIATIONS | 4 |
|---|---|---|---|
| 2 | SIGN | NATURES | 6 |
| 3 | INTE | RODUCTION | 7 |
| 4 | STUI | DY OBJECTIVES AND ENDPOINTS | 7 |
| | 4.1 | Study Objectives | 7 |
| | | 4.1.1 Primary Objective | 7 |
| | | 4.1.2 Secondary Objectives | 7 |
| | 4.2 | Study Endpoints | 8 |
| | | 4.2.1 Primary Endpoints | |
| | | 4.2.2 Secondary Endpoints | |
| | 4.3 | Statistical Hypotheses | 8 |
| 5 | STUI | DY DESIGN | 9 |
| 6 | TIM | E AND EVENTS TABLE | 10 |
| 7 | PLA | NNED ANALYSES | 11 |
| | 7.1 | Interim Analyses | 11 |
| | 7.2 | Final Analysis | 11 |
| | | 7.2.1 Persons responsible for analysis | 11 |
| 8 | SAM | PLE SIZE CONSIDERATIONS | 11 |
| | 8.1 | Sample Size Assumptions | 11 |
| 9 | ANA | LYSIS POPULATIONS | 12 |
| | 9.1 | Analysis Datasets | 12 |
| 10 | TRE | ATMENT COMPARISONS | 13 |
| 11 | GENERAL CONSIDERATIONS FOR DATA ANALYSES | | |
| | 11.1 | Data Display Treatment and Other Subgroup Descriptors | 13 |
| | 11.2 | Conventions for Summary Statistics and Data Displays | 13 |
| 12 | DAT | A HANDLING CONVENTIONS | 14 |
| | 12.1 | Premature Withdrawal and Missing Data | 14 |
| | 12.2 | Derived and Transformed Data | 14 |
| | 12.3 | Assessment Windows | 14 |
| | 12.4 | Values of Potential Clinical Importance | 15 |
| 13 | STUI | DY POPULATION | |
| | 13.1 | Disposition of Patients | |
| | 13.2 | Protocol Deviations | |
| | 13.3 | Baseline Characteristics and Concomitant Medication | |

| | 13.4 | Treatment Compliance | 16 |
|---|---|---|---|
| 14 | SAFI | ETY ANALYSES | 16 |
| | 14.1 | Extent of Exposure | 16 |
| | 14.2 | Adverse Events | 16 |
| | 14.3 | Deaths, Serious Adverse Events and Other Significant Adverse E | vents 17 |
| | 14.4 | Adverse Events Leading to Withdrawal from the Study | 17 |
| | 14.5 | Clinical Laboratory Evaluations | 17 |
| | 14.6 | Other Safety Measures | 17 |
| | | 14.6.1 Vital signs | 17 |
| | | 14.6.2 ECG | 17 |
| 15 | EFFI | CACY ANALYSES | 18 |
| 16 | PHA | RMACOKINETIC ANALYSES | 18 |
| | 16.1 | Pharmacokinetic Concentration Data | 19 |
| 17 | CHA<br>19 | NGES FROM THE PROTOCOL SPECIFIED STATISTICAL | ANALYSIS |
| 18 | REFI | ERENCES | 19 |
| 19 | ATT | ACHMENTS | 20 |
| | 19.1 | Table of Contents for Data Display Specifications | 20 |
| | 19.2 | Data Display Specifications | 24 |
| | | 19.2.1 Table Outlines | 24 |
| | | 19.2.2 Figure Outlines | 35 |
| | | 19.2.3 Listing Outlines | 37 |
| APP | ENDIX | A: SAMPLE PAGE LAYOUT | 46 |

### 1 List of abbreviations

AΕ Adverse Event BEBarrett's esophagus **BMI Body Mass Index** Blood urea nitrogen BUN Cholecystokinin 2 receptor CCK2R CI Confidence Interval Chromogranin A CgA Peak Plasma Concentration  $C_{max}$ Trough Plasma Concentration  $C_{trough}$ Case Report Form CRF Cyclooxygenase-2 COX-2 Clinical Study Report **CSR** CV Coefficient of variance DCAMKL1 Doublecortin- and Ca2+/calmodulin-dependent protein kinase-like protein 1 **ECG** Electrocardiogram Enterochromaffin-like **ECL** Hammersmith Medicines Research HMR HR Heart Rate International Conference on Harmonization **ICH** Immunohistochemistry **IHC** ITT Intent-to-treat LDH Lactase dehydrogenase Medical Dictionary for Regulatory Activities MedDRA Messenger RNA mRNA N Number of patients Number of observations used in analysis N Tumour protein 53 p53 PK Pharmacokinetic(s) PP Per protocol Proton pump inhibitor PPI PR Portion of the ECG from the beginning of the P wave to the beginning of the QRS complex, representing atrioventricular node function. Lower quartile 01 O3 Upper quartile QRS The QRS complex of the ECG reflects the rapid depolarization of the right and left ventricles. qRT-PCR **Ouantitative RT-PCR** QT Portion of the ECG between the onset of the Q wave and the end of the T wave, representing the total time for ventricular depolarization and repolarization. QTc Corrected portion of the ECG between the onset of the Q wave and the end of the T wave, representing the total time for ventricular depolarization and repolarization. OTc interval with Bazett's correction method QTcB QTc interval with Fridericia's correction method **OTcF RBC** Red blood cells

RNAseq RNA sequencing

RR Portion of the ECG between consecutive R waves, representing the

ventricular rate

RT-PCR Reverse transcriptase polymerase chain reaction

SAP Statistical Analysis Plan SD Standard deviation

SGOT/AST Serum glutamic-oxaloacetic transaminase/aspartate amino transferase

SGPT/ALT Serum glutamicpyruvic transaminase/ alanine aminotransferase

TEAE Treatment Emergent Adverse Event

WBC White blood cells

ΔKi67 Change in Ki67 expression

# 2 Signatures

The following persons have read and agreed the content of this Statistical Analysis Plan:

| Stephen Sah<br>Statistics Team Leader, HMR | Signature | Date |
|---|---|---|
| Julian Abrams, MD MS<br>Principal Investigator, Columbia<br>University | Signature | 7-JAN-2019<br>Date |
| Professor Rebecca Fitzgerald<br>Principal Investigator, MRC<br>Cancer Unit | Reduce (174 mol Signature | 21/01/2016) Date |
| Malcolm Boyce<br>Trio Medicines Ltd | Signature Signature | 23 Jan 2019 |

### 3 Introduction

This Statistical Analysis Plan (SAP) is based on the current trial protocol (version 24, 26 April 2018. Where statistical methods differ substantially between this SAP and the protocol, that will be identified in this document.

This SAP describes the datasets and the statistical methods to be used for the reporting and analysis of all data collected during the trial except the efficacy data which will be reported separately. Serum gastrin and plasma CgA data will be included in this SAP.

The randomisation code will not be broken before this SAP is finalised. If a future protocol amendment necessitates a substantial change to the statistical analysis of the trial data, this SAP will be amended accordingly. If, after database lock, additional analyses are required to supplement the planned analyses described in this SAP, those unplanned analyses will not be described in an amended SAP, but they will be identified in the integrated clinical study report (CSR). Any deviations from this SAP will be documented in the CSR.

This SAP has been written in consideration of the following guidelines:

- International Conference on Harmonization (ICH) E9, Guidance for Industry: Statistical Principles for Clinical Trials (ICH E9 1998)<sup>1</sup>; and
- ICH E3, Guidance for Industry: Structure and Content of Clinical Study Reports (ICH E3 1995)<sup>2</sup>.

Statistical analysis will be done using SAS® 9.3 on a Windows PC.

# 4 Study Objectives and Endpoints

# 4.1 Study Objectives

### 4.1.1 Primary Objective

The primary objective of this study is to determine if administration of netazepide (a CCK2R antagonist) to patients with Barrett's esophagus (BE) decreases tissue Ki67 expression, a marker of cellular proliferation.

### 4.1.2 Secondary Objectives

The secondary objectives are to assess the effects of netazepide on:

• biomarkers potentially associated with esophageal adenocarcinoma, in particular, cyclooxygease-2 (COX-2), p53, CCK2R and DCAMKL1; and

• fasting serum gastrin, a marker of gastric acid suppression, and plasma chromogranin A (CgA), a marker of ECL cell hyperplasia.

We also aim to determine whether netazepide is safe in patients with BE.

# 4.2 Study Endpoints

### 4.2.1 Primary Endpoints

Change in Ki67 expression ( $\Delta$ Ki67) between baseline (Visit 2) and the Week 12 visit

### 4.2.2 Secondary Endpoints

- Biomarkers
  - Change from baseline at Week 12 in biomarkers potentially associated with esophageal adenocarcinoma, in particular:
    - Change in CCK2R mRNA levels (measured by qRT-PCR)
    - Change in DCAMKL1 expression (measured by IHC)
    - Change in DCAMKL1 mRNA levels (qRT-PCR)
    - Change in COX-2 mRNA levels (qRT-PCR)
    - Change in p53 expression (IHC)
  - o Gene expression will be measured using RNA-Seq. Further examination of any changes in expression from baseline may be done using qRT-PCR and IHC
  - o Reduction in PPI-induced increase in plasma CgA
  - o Increase in PPI-induced hypergastrinaemia
- Safety
  - Vital signs, ECG, physical examination, laboratory safety tests: blood tests: red blood cells (RBC), haemoglobin, haematocrit, platelets, white blood cells (WBC, differential: neutrophils, bands, lymphocytes, monocytes, eosinophils, basophils), sodium, potassium, magnesium, chloride, bicarbonate, creatinine, serum glucose, blood urea nitrogen (BUN), alkaline phosphatase, lactate dehydrogenase (LDH), serum glutamic-oxaloacetic transaminase/aspartate amino transferase (SGOT/AST), serum glutamicpyruvic transaminase/ alanine aminotransferase (SGPT/ALT), total bilirubin, total protein, albumin, calcium, amylase, lipase; and urine tests: pH, specific gravity, protein, glucose, ketones, blood.
  - Change in histology
- Tolerability: assessment of adverse events.
- Pharmacokinetics: trough and peak concentration of netazepide

### 4.3 Statistical Hypotheses

No formal statistical testing will be done

# 5 Study Design

A randomized, double-blind, placebo-controlled pilot study of netazepide, a cholecystokinin-2 receptor antagonist, in patients with Barrett's esophagus without dysplasia. Patients will take netazepide or placebo for 12 weeks.

There are 2 research sites, Columbia University and the MRC Cancer Unit at the University of Cambridge.

Patients will be randomised (1:1 ratio) to receive either 25 mg netazepide or matching placebo.

### 6 Time and Events Table

| | | ne Testing/<br>y Evaluation | Study to | reatment | Follow-up period |
|---|---|---|---|---|---|
| | Visit 1 <sup>1</sup> | Visit 2 | Week 6<br>visit | Week 12<br>visit | Follow-up |
| Evaluation/ Procedure | Registration | Randomization,<br>& Endoscopy | Week 6 | Week 12 | Follow Up Visit 4 weeks after stopping treatment |
| Informed consent | X | | | | |
| Assess eligibility | X | | | | |
| Central pathology review <sup>2</sup> | X | | | | |
| Medical history | X | | | | |
| Physical exam | X | | | | |
| Vital signs | X | X <sup>5</sup> | X | X | X |
| Height and weight/<br>waist circumference | X | | | | |
| Smoking history | X | | | | |
| Medication history | X | | | | |
| Blood and urine collection for safety tests | X | X <sup>5</sup> | X | X | X |
| Urine pregnancy test <sup>4</sup> | X | X <sup>5</sup> | X | X | X |
| ECG | X | X <sup>5</sup> | X | X | X |
| Blood for YF476 assay <sup>3</sup> | | | X | X | |
| Blood for assay of fasting<br>serum gastrin and plasma<br>CgA, and serum for storage | | X | X | X | X |
| EGD (Upper GI endoscopy) | | X | | X | |
| Biopsies | | X | | X | |
| Concomitant medication assessment | | X | X | X | |
| Dispense study medication | | X | X | | |
| Collect study medication | | | X | X | |
| Compliance assessment | | | X | X | |
| AE assessment | | X | X | X | X |

- 1. There may be up to a 2-week gap between Visits 1 and 2.
- 2. Review of patient's history to obtain histological confirmation of the patient's eligibility to participate in the trial.
- 3. Plasma YF476 assay: patients fast overnight. For the Week 6 and 12 visits, patients bring their container of study medication with them, and take study medication only after collection of blood samples for trough YF476, fasting serum gastrin and CgA levels, and endoscopy (if applicable). Patients stay for 1 h after dosing for collection of a blood sample for peak YF476 level.
- 4. Pre-menopausal women only.
- 5. These tests may be omitted if Visit 2 occurs on the same day as Visit 1.

# 7 Planned Analyses

# 7.1 Interim Analyses

No interim analyses are planned.

# 7.2 Final Analysis

The database will be locked once all patients have completed the study, data have been entered and all queries resolved. The final analysis will be carried out following database lock and unblinding.

### 7.2.1 Persons responsible for analysis

Steven Whaley (HMR) Statistician

Nick Jackson (HMR) SAS Programmer

Jyoti Ambhir (HMR) Data Manager

# 8 Sample Size Considerations

# 8.1 Sample Size Assumptions

Based on preliminary data, a mean baseline Ki67 index of 45–50%, with a common SD of 14-18% was estimated. Assuming a two-sided type I error rate of 0.05, a sample size of 20 (10 per arm) has 98% power to detect a 30% absolute difference in  $\Delta$ Ki67 between the two arms if the common SD is 16%, and 97% power for a 25% difference with a 14% common SD (see Table 1).

| Table 1. Pov | Table 1. Power calculations based on 20 patients (10 per arm) | | |
|---|---|---|---|
| | | $\Delta Ki67_{YF} - \Delta Ki67_{pl}$ | |
| SD | 0.25 | 0.30 | 0.35 |
| 0.14 | 97% | 99% | >99% |
| 0.16 | 91% | 98% | >99% |
| 0.18 | 84% | 94% | 98% |

# 9 Analysis Populations

The following populations will be identified:

Screened Population: All patients screened for the study.

Safety Population: All patients who are randomised and received at least one

dose of the study drug. In this population, treatment will be assigned based upon the treatment patients actually receive regardless of the treatment to which they were randomized.

Intent-to-Treat (ITT) Population: All randomised patients who receive at least one dose of

study medication and had at least one post-baseline

assessment. In this population, treatment will be assigned

based upon the treatment to which subjects were

randomised regardless of which treatment they actually

received.

Per Protocol (PP) Population: All randomized patients who receive at least one dose of

study medication and had at least one post-baseline

assessment and did not have any major protocol deviations.

In all populations (apart from ITT) treatment will be assigned based upon the treatment patients actually receive regardless of the treatment to which they were randomised.

The primary endpoint will be analysed using the ITT population.

### 9.1 Analysis Datasets

All analysis datasets will be based on observed data, except as outlined in Section 12.2.

# 10 Treatment Comparisons

The treatment comparison of interest is active (netazepide) versus placebo.

# 11 General Considerations for Data Analyses

### 11.1 Data Display Treatment and Other Subgroup Descriptors

The sort order for treatment groups will be placebo, then study treatment. When a total column is included, it immediately follows the treatment groups which it aggregates.

Listings of data will be sorted and displayed by treatment group, patient number, and also by date and time if applicable.

The treatment descriptions to be used on all tables and listings are:

### **Treatment Groups**

Placebo

Netazepide 25 mg

# 11.2 Conventions for Summary Statistics and Data Displays

The minimum set of summary statistics for numeric variables will be: n, mean, standard deviation (or standard error), median, minimum, and maximum. 95% confidence intervals will be presented where appropriate for data interpretation.

Categorical data will be summarised in frequency tables with n and percentage. Summaries of a categorical variable will include all recorded values.

The minimum and maximum values will be presented with the same number of decimal places as the raw data collected on the CRF (or to 3 significant figures for derived parameters less than 100 and as integers for values more than 99). The mean and percentiles (e.g. median, Q1, and Q3) will be presented using one additional decimal place. The standard deviation and standard error will be presented using two additional decimal places.

# 12 Data Handling Conventions

### 12.1 Premature Withdrawal and Missing Data

All patients who withdraw prematurely from the study or study drug will be included in the statistical analyses.

If a patient completes the treatment period but has missing data, then this will be made apparent in the patient listings. Missing data will not be imputed except for as outlined in Section 12.2.

If the study is prematurely discontinued, all available data will be listed and a review will be carried out to assess which statistical analyses are still considered appropriate.

Data collected at unscheduled time points during the study will not be used in the summaries or data analyses. They will be included in the listings.

If time information (i.e. hours and/or minutes) for adverse events or concomitant medication is missing, but the day is present, then the time will be calculated in days. If date information is partial or missing, then any derived times (e.g. AE start time from last study medication) will be listed as missing.

### 12.2 Derived and Transformed Data

Baseline will be considered to be the latest value obtained before study drug administration (e.g. Visit 2; or Visit 1 if not recorded elsewhere).

Laboratory data will be reported in standard units. Out-of-range laboratory tests may be repeated. If a test is out-of-range at a baseline timepoint and repeated before dosing, the latest repeat value before dosing will be used as baseline. However, if a test is out-of-range and repeated at any other time during the study, the out-of-range value (not the repeat value) will be included in statistical summaries.

### 12.3 Assessment Windows

There is a +/- 4 day window for clinic visits. Visit 2 can take place on the same day as visit 1, or up to 2 weeks later.

For the safety and ITT populations, all data will be analysed as recorded (regardless of the assessment windows).

### 12.4 Values of Potential Clinical Importance

Laboratory results identified as 'clinically significant' in the CRF will be considered to be potentially clinically important.

QT, QTcB or QTcF > 450 msec and increases in QT, QTcB or QTcF from baseline (Visit 2) of > 30 msec will be considered to be potentially clinically important.

# 13 Study Population

# 13.1 Disposition of Patients

The disposition of all patients in the safety population will be summarised (by site and overall) including number of patients randomised, number completing the study by treatment, and number withdrawn from the study. The number of screen failures will also be summarised and listed.

All patients who withdraw or are withdrawn from the study will be listed by treatment, with the reason for withdrawal

A listing of analysis populations will be provided.

### 13.2 Protocol Deviations

Before closing the database, data listings will be reviewed to identify any significant deviations and determine whether the data should be excluded from any analysis populations.

Major protocol deviations include patients who:

- Entered the study even though they did not satisfy the entry criteria.
- Met the criteria for withdrawal from the study but were not withdrawn.
- Received the wrong treatment or incorrect dose.
- Received an excluded concomitant therapy.
- Received investigational product(s) past the expiration date.
- Had their treatment assignment unblinded.
- Visits outside of assessment windows

### 13.3 Baseline Characteristics and Concomitant Medication

Demographic and baseline characteristics (e.g., vital signs and ECGs) will be listed and summarised.

Patients who take concomitant medication will be listed and summarised.

Proton Pump Inhibitor use data will be listed.

Medical history including history of Barrett's Esophagus data will be listed and summarised

### 13.4 Treatment Compliance

The percentage treatment compliance at each visit will be listed and summarised.

# 14 Safety Analyses

Summaries and listings of safety data will use the safety population.

### 14.1 Extent of Exposure

The dates and times of first and last treatment dosing will be listed to indicate exposure to the study medication.

### 14.2 Adverse Events

Adverse events will be coded using the version of the Medical Dictionary for Regulatory Activities (MedDRA) which is current at the time of database lock (version 20.1 or higher).

All adverse events will be listed.

The number of patients with at least one treatment-emergent adverse event (TEAE) will be tabulated by actual treatment and MedDRA system organ class. A treatment-emergent adverse event is defined as an event emerging during treatment having been absent pretreatment or having worsened relative to pre-treatment<sup>1</sup>.

For each of the following, the number of adverse events and number of patients with adverse events will be summarised by treatment:

- TEAEs by system organ class and preferred term
- Drug-related ("possibly", "probably" or "definitely" as recorded by the Investigator) TEAEs by system organ class and preferred term

Patients with more than one TEAE will be counted only once, at the greatest severity or causality, for each system organ class/preferred term. Multiple TEAEs in a patient will be

counted once per system organ class and preferred term. Adverse events with missing severity and/or causality will be treated as severe and definitely related, respectively.

Summaries will be sorted by system organ class and decreasing total incidence of preferred term.

# 14.3 Deaths, Serious Adverse Events and Other Significant Adverse Events

Deaths and serious adverse events will be listed separately (fatal events separate from non-fatal events). Other significant adverse events, as identified by the investigator in the CRF, will be listed separately.

# 14.4 Adverse Events Leading to Withdrawal from the Study

Adverse events leading to withdrawal will be listed separately.

### 14.5 Clinical Laboratory Evaluations

Data from haematology, clinical chemistry and urinalysis will be summarised by treatment group.

All laboratory values of potential clinical importance will be listed and all related laboratory results (i.e. haematology or clinical chemistry) for patients with values of potential clinical importance will be listed, separately. Frequencies of laboratory values of potential clinical importance will be summarised.

Urinalysis parameters will also be listed.

### 14.6 Other Safety Measures

### 14.6.1 Vital signs

Vital signs evaluation at each planned visit, and change in vital signs from baseline (Visit 2 or Visit 1 if not recorded elsewhere) at each planned post-baseline visit, will be summarised by treatment group.

#### 14.6.2 ECG

QT interval data will be presented using Bazett's (QTcB) and Fridericia's (QTcF) corrections.

ECG data will be summarised by treatment and visit. Differences from baseline (Visit 2) will be summarised by treatment and visit.

The number of patients with a potentially clinically important ECG value will be summarised by actual treatment and visit, giving the numbers of patients with QT, QTcB or QTcF > 450 msec, > 480 msec and > 500 msec, and the numbers of patients with increases in QT, QTcB or QTcF from baseline of > 30 msec and > 60 msec<sup>3</sup>. A supporting listing of all patients with an ECG value of potential clinical importance and a separate listing of ECG findings classified as abnormal by the Investigator will also be provided.

# 15 Efficacy Analyses

Efficacy data (serum gastrin and CgA) will be summarised using the ITT and PP populations. Summaries based on the PP population will only be produced if there is a difference between the ITT and PP populations

Serum gastrin and plasma CgA data at each planned visit, and change in Serum gastrin and plasma CgA from baseline at each planned post-baseline visit, will be summarised by treatment group and visit. Individual values will be presented by patient

Mean profile plots for serum gastrin and CgA will also be produced. Each plot will contain all results for all subjects in the active and placebo arms

# 16 Pharmacokinetic Analyses

Analytics Services International Ltd. will measure the plasma concentrations of netazepide. The pharmacokinetic analysis will be done by HMR.

PK data will be summarised using the safety population for patients who received netazepide 25 mg.

For all variables N (number of patients receiving the treatment in the population), n (number of observations), arithmetic mean, median, minimum, maximum, SD, %CV, and the 95% confidence interval for the arithmetic mean will be provided.

### 16.1 Pharmacokinetic Concentration Data

The peak  $(C_{max})$  and trough  $(C_{trough})$  plasma concentration will be listed, presented graphically and summarised by treatment.

We will produce scatterplots to examine the relationship between peak PK concentrations and plasma CgA concentration or serum gastrin concentration.

# 17 Changes from the Protocol Specified Statistical Analysis

After the study was submitted to the regulatory authorities and ethics committee the following changes were made to the analyses:

 Section 13.1 Analysis Sets of the protocol states "The pharmacokinetic analysis set will include all patients who receive at least one dose of study medication, and yield at least one plasma concentration for netazepide." This definition is not included in the SAP as the population is not required.

### 18 References

- 1. International Conference on Harmonization, 1998. Statistical Principles for Clinical Trials ICH Harmonised Tripartite Guideline. Guidance for Industry, E9, FDA federal register, Vol 63, 1998, p49583. Available at: http://www.fda.gov/cder/guidance.
- 2. International Conference on Harmonization, 1995. Structure and Content of Clinical Study Reports ICH Harmonised Tripartite Guideline. Guidance for Industry, E3, FDA federal register, Vol 61, 1996, p37320. Available at: http://www.fda.gov/cder/guidance.
- 3. International Conference on Harmonisation, 2005. Clinical Evaluation of QT/QTc Interval Prolongation and Proarrhythmic Potential for Non-Antiarrhythmic Drugs. Concept paper, Guidance for Industry, E14, Center for Drug Evaluation and Research (CDER). Available at: http://www.fda.gov/cder/guidance/6922fnl.htm.

# 19 ATTACHMENTS

# 19.1 Table of Contents for Data Display Specifications

For overall page layout refer to Appendix B.

The numbering in the tables below will take precedence over the numbering in the shells.

The following tables and figures will be produced (templates provided in Section 19.2.1 and 19.2.2):

| Table | Description | Population | Source<br>Listing | Template (Shells below) |
|---|---|---|---|---|
| 10.1 | Summary of patient disposition | Safety | 16.2.1.2 | <u>T_SD1</u> |
| | | | 16.2.3.1 | |
| 10.2.1 | Summary of concomitant medications | Safety | 16.2.4.2 | <u>T_CM1</u> |
| 10.2.2 | Summary of medical history: barrett's esophagus | Safety | 16.2.4.3 | <u>T_MH1</u> |
| 10.2.3 | Summary of treatment compliance | Safety | 16.2.5.1 | T_COMP1 |
| 14.1 | DEMOGRAPHIC DATA | | | |
| 14.1 | Summary of demographic characteristics | Safety | 16.2.4 | T DM1 |
| 14.2 | PHARMACOKINETIC and EFFICACY | | | |
| 14.2.1 | Summary of netazepide plasma peak and trough concentration data | Safety | 16.2.6.1 | <u>T_PK1</u> |
| 14.2.2.1 | Summary of serum gastrin and plasma CgA data (ITT) | ITT | 16.2.6.2 | T EG2 |
| 14.2.2.2* | Summary of serum gastrin and plasma CgA data (PP) | PP | 16.2.6.2 | T_EG2 |
| 14.3 | SAFETY DATA | | | |
| 14.3.1.1 | Summary of treatment-emergent adverse events | Safety | 16.2.7.1 | T_AE1 |
| 14.3.1.2 | Summary of drug-related treatment-emergent adverse events | Safety | 16.2.7.1 | <u>T_AE1</u> |
| 14.3.2.1 | Listing of fatal adverse events | Safety | 16.2.7.1 | L_AE1_PG |
| 14.3.2.2 | Listing of non-fatal serious adverse events | Safety | 16.2.7.1 | L_AE1_PG |
| 14.3.2.3 | Listing of other significant adverse events | Safety | 16.2.7.1 | L_AE1_PG |
| 14.3.3 | Narratives of deaths, other serious and significant adverse events | Safety | - | - |
| 14.3.4 | Summary of laboratory values of potential clinical importance | Safety | 16.2.8.1, | <u>T_LB1</u> |
| | | | 16.2.8.3 | |
| 14.3.5.1 | Summary of chemistry laboratory values | Safety | 16.4 | <u>T_LB2</u> |
| 14.3.5.2 | Summary of haematology laboratory values | Safety | 16.4 | <u>T_LB2</u> |
| 14.3.5.3 | Summary of urinalysis results | Safety | 16.4 | T_UR1 |
| 14.3.6.1 | Summary of vital signs | Safety | 16.4 | <u>T_VS1</u> |
| 14.3.7.1 | Summary of ECG values | Safety | 16.4 | T_EG2 |
| 14.3.7.2 | Summary of ECG values and changes in ECG values of potential clinical importance | Safety | 16.4 | T_EG3 |

| Figure | Description | Population | Source<br>Listing | Template (Shells below) |
|---|---|---|---|---|
| 14.3 | SAFETY AND EFFICACY DATA | | | |
| 14.3.1 | Individual netazepide plasma concentration plots | Safety | 16.2.6.1 | F PK1 |
| 14.3.2.1.1 | Mean $\pm$ SD serum gastrin – time plot (ITT) | ITT | 16.2.6.2 | F PK4 |
| 14.3.2.1.2* | Mean $\pm$ SD serum gastrin – time plot (PP) | PP | 16.2.6.2 | F PK4 |
| 14.3.2.2.1 | Mean $\pm$ SD plasma CgA – time plot (ITT) | ITT | 16.2.6.2 | F PK4 |
| 14.3.2.2.2* | Mean $\pm$ SD plasma CgA – time plot (PP) | PP | 16.2.6.2 | F PK4 |

<sup>\*</sup>Only produce if there is a difference between ITT and PP populations

The following listings will be produced (templates found in section 19.2.3)

| Listing | Description | Template (Shells<br>below) |
|---|---|---|
| 16.2.1 | Study dates & disposition of patients | , |
| 16.2.1.1 | Listing of study dates | L SD1 PG |
| 16.2.1.2 | Listing of reasons for withdrawal | L SD2 PG |
| 16.2.1.3 | Listing of screen failures | L SD3 PG |
| 16.2.2 | Protocol deviations | |
| 16.2.2.1 | Listing of patients with inclusion/exclusion criteria deviations | L DV1 PG |
| 16.2.2.2 | Listing of patients with other protocol deviations | L_DV2_PG |
| 16.2.3 | Analysis sets, including patients excluded from analysis | |
| 16.2.3.1 | Listing of analysis populations | L AN1 PG |
| 16.2.4 | Demographic data & concomitant medication | |
| 16.2.4.1 | Listing of demographic characteristics | L DM1 PG |
| 16.2.4.2 | Listing of concomitant medications | L CM1 PG |
| 16.2.4.3 | Listing of medical history: barrett's esophagus | L_MH1_PG |
| 16.2.4.4 | Listing of proton pump inhibitor use | L PP1 PG |

| Listing | Description | Template (Shells below) |
|---|---|---|
| 16.2.5 | Study drug administration | · |
| 16.2.5.1 | Listing of study drug administration and treatment compliance | L EX PG |
| 16.2.6 | Pharmacokinetic and Efficacy data | |
| 16.2.6.1 | Listing of netazepide plasma pharmacokinetic data | L PK1 PG |
| 16.2.6.2 | Listing of serum gastrin and plasma CgA data | L_PK4_PG |
| 16.2.7 | Adverse events | |
| 16.2.7.1 | Listing of all adverse events | L AE1 PG |
| 16.2.7.2 | Listing of serious adverse events | L_AE1_PG |
| 16.2.7.3 | Listing of adverse events leading to withdrawal from study | L AE1 PG |
| 16.2.8 | Laboratory values | |
| 16.2.8.1 | Listing of clinical chemistry abnormalities of potential clinical importance | L LB1 PG |
| 16.2.8.2 | Listing of all clinical chemistry laboratory data for patients with PCI abnormalities | L_LB2_PG |
| 16.2.8.3 | Listing of haematology abnormalities of potential clinical importance | L_LB1_PG |
| 16.2.8.4 | Listing of all haematology laboratory data for patients with PCI abnormalities | L_LB2_PG |
| 16.2.8.5 | Listing of urinalysis results | |
| 16.2.9 | ECG variables | |
| 16.2.9.1 | Listing of ECG values of potential clinical importance | L_EG1_PG |
| 16.2.9.2 | Listing of abnormal ECG findings | L EG2 PG |

Complete listings of all data collected in this study will also be produced.

# 19.2 Data Display Specifications

# 19.2.1 Table Outlines

### Template T\_SD1

Table 10.1 Summary of Patient Disposition

| Population | Status | Reason for Withdrawal | | Treatment 1 | Etc | | All Patients | |
|---|---|---|---|---|---|---|---|---|
| | | | Columbia | Cambridge | All Sites | Columbia | Cambridge | All Sites |
| | | | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Screened | Included | | XX | XX | XX | XX | XX | XX |
| Safety | Included | | XX | XX | XX | XX | XX | XX |
| | Completed | | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx(xx) | xx (xx) |
| | Withdrawn | | | | | | | |
| | | Death | xx(xx) | xx(xx) | xx (xx) | xx(xx) | xx(xx) | xx(xx) |
| | | Adverse Events | xx(xx) | xx(xx) | xx (xx) | xx(xx) | xx(xx) | xx (xx) |
| | | Withdrawal by patient | xx(xx) | xx (xx) | xx (xx) | xx (xx) | xx(xx) | xx (xx) |
| | | Physician decision | xx(xx) | xx(xx) | xx (xx) | xx(xx) | xx(xx) | xx(xx) |
| | | Protocol violation | xx(xx) | xx(xx) | xx (xx) | xx(xx) | xx(xx) | xx(xx) |
| | | Pregnancy | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx(xx) | xx(xx) |
| | | Study terminated by | xx(xx) | xx(xx) | xx (xx) | xx(xx) | xx(xx) | xx(xx) |
| | | Sponsor | | | | | | |
| | | Lost to follow-up | | | | | | |
| | | Other | xx(xx) | xx(xx) | xx (xx) | xx (xx) | xx(xx) | xx (xx) |
| Intent to Treat | Included | | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| | Completed | | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| | Withdrawn | | | | | | | |
| | | Death | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| | | Adverse Events | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| | | Withdrawal by patient | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| | | Physician decision | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| | | Protocol violation | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) |

| | | Pregnancy | xx(xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx(xx) |
|---|---|---|---|---|---|---|---|---|
| | | Study terminated by | xx(xx) | xx(xx) | xx (xx) | xx (xx) | xx(xx) | xx(xx) |
| | | Sponsor | | | | | | |
| | | Lost to follow-up | | | | | | |
| | | Other | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx(xx) |
| Per Protocol | Included | | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) |

Source: Listing 16.2.xx

Programming notes: Continued with all treatment groups

### Template T\_CM1

Table 10.2.2 Summary of Concomitant Medications

| Generic Term | | ment 1<br>=xx) | Treatment 2<br>(N=xx) | |
|----------------|---|----------------|-----------------------|---|
| | n | % | n | % |
| Any medication | | • | | • |
| Medication 1 | | | | |
| Medication 2 | | | | |
| Medication 3 | | | | |
| Medication 4 | | | | |

Source: Listing 16.2.xx

Programming notes: Continued with all treatment groups

### Template T\_COMP1

Table 10.2.2 Summary of Treatment Compliance

| Variable | Treatment | Visit | n | Mean | SD | Median | Min | Max |
|---|---|---|---|---|---|---|---|---|
| Compliance (%) | Treatment 1 (N=xx) | | | | | | | |

Programming notes: Continued with all treatment groups

### Template T\_MH1

Table 10.2.2 Summary of Medical History: Barrett's Esophagus

| | Treatr | Treatment 2<br>(N=xx) | | |
|---------------------|--------|-----------------------|---|---|
| Barrett's mucosa | (N= | | | |
| | n | % | n | % |
| Circumferential | | | | |
| Non-circumferential | | | | |

### Template T\_DM1

Table 14.1 Summary of Demographic Characteristics

| Variable | Statistics | Screen Failures | Treatment 1 | Treatment 2 | Etc | All Treated Patients |
|---|---|---|---|---|---|---|
| | | (N=xx) | (N=xx) | (N=xx) | | (N=xx) |
| Age (y) | n | | | | | |
| | Mean | | | | | |
| | SD | | | | | |
| | Median | | | | | |
| | Min | | | | | |
| | Max | | | | | |
| Gender | N | | | | | |
| | Female | | | | | |
| | Male | | | | | |
| Race | American Indian | | | | | |
| | Asian/ Pacific Islander | | | | | |
| | Black | | | | | |
| | Hispanic | | | | | |
| | White | | | | | |
| | Other | | | | | |
| Height (cm) | n | | | | | |
| | Mean | | | | | |
| | SD | | | | | |
| | Median | | | | | |
| | Min | | | | | |
| | Max | | | | | |
| Weight (kg) | n | | | | | |
| | Mean | | | | | |
| | SD | | | | | |
| | Median | | | | | |
| | Min | | | | | |
| | Max | | | | | |

| Variable | Statistics | Screen Failures<br>(N=xx) | Treatment 1<br>(N=xx) | Treatment 2<br>(N=xx) | Etc | All Treated Patients<br>(N=xx) |
|---|---|---|---|---|---|---|
| BMI (kg/m2) | n | | | | | |
| | Mean | | | | | |
| | SD | | | | | |
| | Median | | | | | |
| | Min | | | | | |
| | Max | | | | | |
| Waist | n | | | | | |
| circumference | Mean | | | | | |
| (cm) | SD | | | | | |
| | Median | | | | | |
| | Min | | | | | |
| | Max | | | | | |
| Cigarettes* | n | | | | | |
| (daily) | Mean | | | | | |
| | SD | | | | | |
| | Median | | | | | |
| | Min | | | | | |
| | Max | | | | | |
| Alcohol* | n | | | | | |
| (units/week) | Mean | | | | | |
| | SD | | | | | |
| | Median | | | | | |
| | Min | | | | | |
| | Max | | | | | |

<sup>\*</sup>includes only those patients who smoke/drink alcohol

Source: Listing 16.2.xx

Programming notes: Continued with all treatment groups and additional demographic characteristics

### Template T\_AE1

Table 14.3.3.xx Summary of Treatment-Emergent Adverse Events

| | | Treatment 1 (N=xx) | Treatment 2 (N=xx) Etc |
|---|---|---|---|
| System Organ Class | Preferred Term | n (%) | n (%) |
| Number of patients with AEs | | x (xx.x) | x (xx.x) |
| Gastrointestinal disorders | Total number of patients | x (xx.x) | x (xx.x) |
| | Abdominal discomfort | x (xx.x) [xx] | x (xx.x) [xx] |
| | Abdominal pain | x (xx.x) [xx] | x (xx.x) [xx] |
| | $\downarrow$ | | |
| Nervous system disorders | Total number of patients | | |
| | Dizziness | | |
| | Headache | | |
| | $\downarrow$ | | |
| $\downarrow$ | $\downarrow$ | | |

n = number of patients (patients with ≥1 adverse event are counted only once per system organ class and preferred term)

[] = number of TEAEs

Based on MedDRA version xx.x

Source: Listing 16.2.xx

Programming notes: Continued with all treatment groups

SOCs and PTs are sorted in decreasing order of frequency

Presented for all applicable MedDRA system organ classes and terms.

### Template T\_LB1

Table 14.3.4.xx Summary of Laboratory Values of Potential Clinical Importance

| Laboratory Test (units) | Treatment | Visit | n (%) |
|-------------------------|--------------------|-------|-------|
| | Treatment 1 (N=xx) | | |

Source: Listing 16.2.xx

Programming notes: Continued with all tests, treatment groups and time points. n = total number of results for that parameter

### Template T\_LB2

Table 14.3.5.xx Summary of Chemistry Laboratory Values

| | | | | | | | | | Change from Baseline | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Laboratory Test | | | | | | | | | | | | | | |
| (units) | Treatment | Visit | n | Mean | SD | Median | Min | Max | n | Mean | SD | Median | Min | Max |
| | Treatment 1 (N=xx) | | | | | | | | | | | | | |

Source: Listing 16.2.xx

Programming notes: Continued with all treatments and time points For Ki67 Expression data exclude first column

### Template T\_UR1

Table 14.3.5.xx Summary of Urinalysis Results

| | | | Treatment 1 | L (N=xx) | Treatment 2 (N=xx) | |
|---|---|---|---|---|---|---|
| Laboratory Test | Visit | Result | n | % | n | % |
| | Time 1 | Positive | Х | х | | |
| | | Negative | Х | Χ | | |
| | | Not Done | х | | | |
| | Time 2 | Positive | | | | |
| | | Negative | | | | |
| | | Not Done | | | | |

Source: Listing 16.2.xx

Programming notes: Results recorded as received, e.g. Negative, Trace, etc; urine pH summarized as <5, 5-8, >8

Continued with all treatment groups and time points. The n's sum to N but the calculated percentages exclude Not Done.

### Template T\_VS1

Table 14.3.6.xx Summary of Vital Signs

| | | | | | | | | | Change from Baseline | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Variable (units) | Treatment | Visit | n | Mean | SD | Median | Min | Max | n | Mean | SD | Median Min | Max |
| Systolic BP (mmHg) | Treatment 1 (N=xx) | | | | | | | | | | | | |

Source: Listing 16.2.xx

Programming notes: Continued with all variables, treatments and time points

### Template T\_EG2

Table 14.3.7.xx Summary of ECG Values

| | | | | | | | | | | Cl | nange | from Baseli | ne | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Variable (units) | Treatment | Visit | n | Mean | SD | Median | Min | Max | n | Mean | SD | Median | Min | Max |
| Heart Rate (bpm) | Treatment 1 (N=xx) | | | | | | | | | | | | | |
| | Treatment 2 (N=xx) | | | | | | | | | | | | | |
| PR Interval (msec) | Treatment 1 (N=xx) | | | | | | | | | | | | | |
| | Treatment 2 (N=xx) | | | | | | | | | | | | | |

Source: Listing 16.2.xx

Programming notes: Continued with all treatment groups and time points

Do not summarise RR or QRS axis

Template T\_EG3

Table 14.3.7.xx Summary of ECG Values and Changes in ECG Values of Potential Clinical Importance

| | · | | · | | | | | | >30-6 | 0 msec | >60 | msec |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | 451 – 48 | 0 msec | 481 – 5 | 00 msec | > 500 msec | | Incr | ease | Incr | ease |
| Variable | Treatment | Visit | n | % | n | % | n | % | n | % | n | % |
| QT interval | Treatment 1 | Time 1 | | | | | | | | | | |
| | (N=xx) | Time 2 | | | | | | | | | | |
| | | Time 3 | | | | | | | | | | |
| | Treatment 2 | Time 1 | | | | | | | | | | |
| | (N=xx) | Time 2 | | | | | | | | | | |
| | | Time 3 | | | | | | | | | | |
| QTcB interval | Treatment 1 | Time 1 | | | | | | | | | | |
| | (N=xx) | Time 2 | | | | | | | | | | |
| | | Time 3 | | | | | | | | | | |
| | Treatment 2 | Time 1 | | | | | | | | | | |
| | (N=xx) | Time 2 | | | | | | | | | | |
| | | Time 3 | | | | | | | | | | |
| QTcF interval | Treatment 1 | Time 1 | | | | | | | | | | |
| | (N=xx) | Time 2 | | | | | | | | | | |
| | | Time 3 | | | | | | | | | | |

Source: Listing 16.2.xx

Programming notes: Continued with all treatments and time points. n = total number of results for that parameter

Template T\_PK1

Table 14.2.xx Summary of Netazepide Plasma Pharmacokinetic Peak and Trough Concentration Data

| Measurement | Treatment | Visit | n | Mean | SD | %CVb | Median | Min | Max | Geom | 95% CI |
|---|---|---|---|---|---|---|---|---|---|---|---|
| (units) | | | | | | | | | | Mean | (Lower,Upper) |
| Peak | Treatment 1 | Visit 3 | x | xxxx.x | | xx.x | xxxx.x | XXXX | xxxx | | (xxxx.x,xxxx.x) |
| | (N=xx) | Visit 4 | x | XXXX.X | XX.XX | XX.X | XXXX.X | XXXX | XXXX | | (xxxx.x,xxxx.x)<br>(xxxx.x,xxxx.x) |
| Trough | Treatment 1 | Visit 3 | х | xxxx.x | | xx.x | xxxx.x | xxxx | xxxx | | (voucins) |
| | (N=xx) | Visit 4 | х | XXXX.X | XX.XX | XX.X | xxxx.x | XXXX | XXXX | | |

Source: Listing 16.2.xx

# 19.2.2 Figure Outlines

### Template F\_PK1

Figure 14.3.1 Individual Netazepide Plasma Concentration-Time Plots



Programming notes: All patients will be displayed in the same graph on one page.

### Template F\_PK4

Figure 14.3.4 Mean ± SD serum gastrin – time plot (ITT)



### 19.2.3 Listing Outlines

#### Template L\_SD1\_PG

Listing 16.2.x.xx Listing of Study Dates

Treatment Patient Visit 1 Visit 2 Week 6 Visit Week 12 Visit Follow Up

Programming notes: Lists dates for screening, each dosing period and follow up

For crossover studies use Sequence instead of Treatment

### Template L\_SD2\_PG

Listing 16.2.x.xx Listing of Reasons for Withdrawal

Date of Study
Treatment Patient Withdrawal Day Reason

Programming notes: Reason for withdrawal is concatenation of reason and details

### Template L\_SD3\_PG

Listing 16.2.x.xx Listing of Screen Failures

Date of

Patient Screen Failure Failure Category Details

### Template L\_DV1\_PG

Listing 16.2.x.xx Listing of Patients with Inclusion/Exclusion Criteria Deviations

| | Treatment | Patient | Туре | Criterion |
|---|-----------|---------|-----------|-----------|
| _ | | | Inclusion | |
| | | | Exclusion | |

### Template L\_DV2\_PG

Listing 16.2.x.xx Listing of Patients with Other Protocol Deviations

| Treatment | Patient | Protocol Deviation |
|--------------|---------|-----------------------|
| 11 Cutilicit | rationt | 1 TO LOCOL DE VIALION |

### Template L\_AN1\_PG

Listing 16.2.x.xx Listing of Analysis Populations

| | | Screened | Safety | | |
|---|---|---|---|---|---|
| Treatment | Patient | Population | Population | ITT Population | PP Population |

### Template L\_DM1\_PG

Listing 16.2.x.xx Listing of Demographic Characteristics

| | | | | Age | | | | Height | Weight | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | Patient | Date of visit | Date of birth | (y) | Gender | Race | Ethnic origin | (cm) | (kg) | BMI (kg/m2) | Etc (units) |
| Treatme | nt 1 | | | | | | | | | | |
| <b>\</b> | | | | | | | | | | | |
| Programming n | otes: A | by-patient listing of | f demographic char | acteristic | s including: | | | | | | |
| | | Treatment | | | | | | | | | |
| | | Patient | | | | | | | | | |
| | | Date of visit | | | | | | | | | |
| | | Date of birth | | | | | | | | | |
| | | Age | | | | | | | | | |
| | | Gender | | | | | | | | | |
| | | Race / Ethnic C | Origin | | | | | | | | |
| | | Height (if collec | cted only once duri | ng the stu | dy) | | | | | | |
| | | Weight (if colle | cted only once duri | ng the stu | dy) | | | | | | |
| | | Smoking Histor | y | | | | | | | | |
| | | Alcohol Consur | nption | | | | | | | | |
| | | Additional stud | y-specific demogra | phy chara | cteristics incli | ided on the CRI | Ţ. | | | | |

### Template L\_CM1\_PG

Listing 16.2.x.xx Listing of Concomitant Medications

| | | Drug Name/ | Dose/ | Date/time Started/ | Time Since Last | Started Pre- | Ongoing |
|---|---|---|---|---|---|---|---|
| Treatment | Patient | Indication | Freq/Route | Date Stopped | Dose | Trial? | Medication? |

Programming notes: Include dose and units (e.g. 5 mg)/Freq/Route

### Template L\_PP1\_PG

Listing 16.2.x.xx Listing of Proton Pump Inhibitor Use

| | | | | | How often | | | |
|---|---|---|---|---|---|---|---|---|
| | | | | | does the | | | |
| | | | Is patient taking | Have they been | patient | | | |
| | | | proton pump | taking it for at least | take the | Generic | | |
| Treatment | Patient | Date/Time | inhibitor? | 12 months? | PPI? | name | Dose | Date Started |
| Treatment 1 | 1001 | 0114N2002 | Ves | Ves | Once daily | | | |

### Template L\_MH1

Listing 16.2.x.xx Listing of Medical History: Barrett's Esophagus

| | | | | Most | Intestinal | | Maximum |
|---|---|---|---|---|---|---|---|
| | | | | recent | metaplasia | Is Barrett's | measurement |
| | | | | endoscopy | and no | mucosa | of Barrett's |
| Treatment | Patient | Date/Time | Endoscopy | date | dysplasia | circumferential | mucosa (cm) |
| Treatment 1 | 1001 | 01JAN2002 | Yes | | Yes | Yes | |

### Template L\_EX1\_PG

Listing 16.2.x.xx Listing of Study Drug Administration

| | | | | Dur- | | | | | Visit 3 | Visit 4 |
|---|---|---|---|---|---|---|---|---|---|---|
| | | Start Date/ | Stop Date/ | ation | | Dose | Formulation/ | | Compliance | Compliance |
| Treatment | Patient | Start Time of Dose | Stop Time of Dose | (days) | Dose | Unit | Route | Frequency | (%) | (%) |
| Treatment 1 | 1001 | 01JAN2002 | 15FEB2002 | 46 | 25 | mg | Tablet/ | 2xday | | |
| | | 23:59 | 15:30 | | | | Oral | | | |

### Template L\_AE1\_PG

Listing 16.2.x.xx Listing of All Adverse Events

| | | | Outcome/ | | | Frequency/ | Related to Study |
|---|---|---|---|---|---|---|---|
| | | System Organ Class / | Onset Date/Time/ | | Severity/ | Action Taken (1)/ | Drug/ |
| | | Preferred Term/ | Resolved Date/Time/ | Time Since Last | Serious/ | Other Action | Treatment |
| Treatment | Patient | Verbatim Text | Duration | Dose | Withdrawal | Taken | Emergent? |
| Treatment 1 | 1001 | Gastrointestinal Disorders / | Resolved/ | 10d 7h 3m | Mild/ | Intermittent/ Dose | Possibly/ |
| | | Intestinal Spasm / | 24SEP2003 13:05/ | | No/ | not changed/ | Yes |
| | | Entero-spasm | 27OCT2003 7:50/ | | Yes | None | |
| | | | 34d 4h 5m | | | | |

<sup>(1)</sup> Action Taken with Study Treatment

Programming notes: For the listing of "other significant AEs" include (from ICH E3) AEs leading to withdrawal, AEs leading to dose reduction (including drug withdrawn, interrupted, reduced or similar) and AEs with AEOSE=Y. If AEOSE has not been collected then use "Otherwise significant" in the CRF.

Template L\_LB1\_PG

Listing 16.2.x.xx Listing of clinical chemistry abnormalities of potential clinical importance

| | | | Planned | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | | Relative | | Study | | | Clinically |
| Treatment | Subject | Laboratory test (units) | Time | Date/Time | Day | Value | Reference Interval | Significant? |
| Treatment 1 | 1001 | Alk Phos (U/L) | Time 1 | 01JAN2002 | -1 | 64.00 | 32.0 - 92.0 | Υ |
| | | | | 13:34 | | | | |
| | | | Time 2 | 01APR2002 | 85 | 84.00 | 32.0 - 92.0 | Υ |
| | | | | 07:22 | | | | |
| | | ALT (U/L) | Time 1 | 01JAN2002 | -1 | 29.00 | 10.0 - 40.0 | Υ |
| | | | | 18:56 | | | | |
| | | | Time 2 | 01APR2002 | 85 | 70.00 | 10.0- 40.0 | Υ |
| | | | | 09:22 | | | | |

Programming notes: Lists only Laboratory results identified as 'clinically significant' in the CRF

### Template L\_LB2\_PG

Listing 16.2.x.xx Listing of all clinical chemistry laboratory data for subjects with PCI abnormalities

| | | Planned<br>Relative | | Alkaline Phos | phatase (IU/L) | | o Transferase<br>/L) | Aspartate Amin | | Total Bilirubin (UMOL/L) |
|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | Subject | Time | Date/Time | Result | | Result | | Result | | Result |
| | | | | xx* | | x.xx | | | | |
| | | Planned | | | | | | | | |
| | Relative | | | Chloride (MMOL/L) | | Glucose (MMOL/L) | | Potassium (MMOL/L) | | Sodium (MMOL/L) |
| Treatment | Subject Time | | Date/Time | Result | Result | | | Result | | Result |
| | | | Planned | | | | | | | |
| | | | Relative | | Calcium ( | (MMOL/L) | Creatinin | e (UMOL/L) | | Etc. |
| | Treatm | nent Subject | : Time | Date/Time | Result | | Result | | Result | |

<sup>\*</sup> Value of potential clinical significance

Programming notes:

Lists only subjects identified as 'clinically significant' in the CRF Include all parameters for the study following the order from the lab report (above is a guide only)

### Template L\_EG1\_PG

Listing 16.2.x.xx Listing of ECG Values of Potential Clinical Importance

| | | | | | | | | QT Int. | QT Int. (msec) QT | | (msec) | QTcF ( | (msec) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | Heart | | QRS | QRS | | Change | | Change | | Change |
| | | Planned | | Rate | PR Int. | Dur. | Axis | | from | | from | | from |
| Treatment | Patient | ient Relative Time Date/Time | | (bpm) | (msec) | (msec) | (deg) | Observed | Baseline | Observed | Baseline | Observed | Baseline |
| | | 24 H | 26SEP2012:09:57 | 63 | 148 | 78 | 50 | 390 | 32.7 * | 399 | -27.7 | 396 | -6.5 |

Programming notes: Do not list RR

### Template L\_EG2\_PG

Listing 16.2.x.xx Listing of Abnormal ECG Findings

| Planned Relative | | | | Comment on Clinical | |
|---|---|---|---|---|---|
| Treatment | Patient | Time | Date/Time | ECG Finding | Significance |

Programming notes: Lists only values with Normal variant='No' or with comment on ECG result

ECG Finding contains Physician's Opinion from CRF and relates to whole trace (not individual parameters), e.g. Normal, Abnormal - NCS or Abnormal - CS

<sup>\*</sup> Value of potential clinical importance

### Template L\_PK1\_PG

Listing 16.2.6.xx Listing of Netazepide Plasma Pharmacokinetic Parameters

| | | | Planned | Concentration (units) | |
|---|---|---|---|---|---|
| Treatment | Patient | Date | <b>Relative Time</b> | Peak (C <sub>max</sub> ) | Trough (C <sub>min</sub> ) |

### Template L\_PK4\_PG

Listing 16.2.6.xx Listing of serum gastrin and plasma CgA data

| | Planned | | | | |
|-----------|---------|------|---------------|---------------|-----------|
| Treatment | Patient | Date | Relative Time | Serum Gastrin | Plasma Cg |

# **Appendix A: Sample Page Layout**

| Trio Medicines Ltd : T-016 | Page x of y* | |
|---|---|---|
| Population: [Pop] | | |
| | Table [number] [title] | |
| | Column headers | • |
| | Main body of output | |
| | Source: Listing [16.2.xx] | |
| Footnotes about the table or list | ing text go here. | |
| Program: [Prog Name] Produced By:[Username] | [Date] | HMR 10-505 |

Font size will be Arial 9.5pt. The following margins will be used: Left: 1", Right: 1", Top: 1", Bottom: 1"

<sup>\*</sup>y = last page of individual output